CLINICAL TRIAL: NCT02733406
Title: The Effect of Target Controlled Infusion as Opposed to Velocity Controlled Infusion on Hypotension at Induction of Total Intravenous Anaesthesia
Brief Title: Hypotensive Effect of Anaesthesia With TCI
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Joakim Johansson, Dr Joakim Johansson, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TCI hypotension TIVA
Record Dates: First submitted 2016-03-21; First posted 2016-04-11 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Blood Pressure; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Target Controlled Infusion (Other): This group of patients will have their anaesthesia induced with Target Controlled Infusion (TCI)
  Interventions: Other: Target Controlled Infusion
- Velocity Controlled Infusion (Other): This group of patients will have their anaesthesia induced with Velocity Controlled Infusion (VCI)
  Interventions: Other: Velocity Controlled Infusion

INTERVENTIONS:
Other: Target Controlled Infusion
  Arms: Target Controlled Infusion
Other: Velocity Controlled Infusion
  Arms: Velocity Controlled Infusion

SUMMARY:
Hypotension will often complicate induction of anaesthesia. The investigators want to test the hypothesis that Target Controlled Infusion, as opposed to Velocity Controlled Infusion, leads to less degree of hypotension.

DETAILED DESCRIPTION:
Severe hypotension may be a serious complication to induction of anaesthesia. The patients preoperative clinical circulatory status will help define the risks of such a side-effect. A patient with a preexisting heart condition will be at increased risk for morbidity/mortality in relation to anaesthesia induction.

Total intravenous anaesthesia may be delivered by two different approaches. The old way where the drug (Propofol and/or Remifentanil) is delivered in a velocity (mg/kg x hour or microg/ kg x min) specified by the anaesthetist. Hereafter called Velocity Controlled Infusion (VCI). At induction, to get effect of the drug, a high infusion rate is desired. A high infusion rate is associated with increased risks of hypotension if it is not adjusted in accordance with the current circulatory status of the patient. A failure to adjust may be futile for the patient. Therefore, induction takes some time because infusion rate is set within a relatively safe range. After a few minutes, once airway control is achieved, the infusion rate must be adjusted down to avoid hypotension.

There is a more modern way of adjusting the infusion rate, the so called Target Controlled Infusion. With this approach, the pump delivering the drug will help the anaesthetist to select the appropriate infusion rate for any given situation. The anaesthetist selects a preferred concentration of the drug at the target, that is in the circulation. The pump then administrates the drug, first at high rate and then at lower rate, taking into account the patients age, weight and sex and the preferred target concentration.

It is possible that this help from the machine is associated with less risk for hypotension at anaesthesia induction. If this is so it would have an impact on which of TCI and VCI that would be the best choice of anaesthesia. This would have special impact when giving anaesthesia to patients with a heart condition.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for anaesthesia at Östersunds Hospital

* ASA class I-II

Exclusion Criteria:

* On beforehand decision to start continous delivery of blood pressure increasing drug at induction.
* Any contraindication to Total Intravenous Anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Hypotension | 20 minutes
  Relative maximal decrease of blood pressure (in mmHg) by anaesthesia induction (%)

SECONDARY OUTCOMES:
Pharmacological measures to increase blood pressure | 20 minutes
  Number of doses of drug to increase blood pressure
Drug consumption | From the start of anaesthesia induction to the time of airway control (Laryngeal airway working in place of tracheal tube working in place).
  Amount (milligram) of Propofol delivered and amount (mikrogram) of Remifentanil delivered.
PONV (Postoperative Nausea and Vomiting) | From end of anaesthesia to 2 hours or when leaving the PostAnaesthesia Care Unit
  Dose and name of any drug given to reduce PONV at any time defined above (in addition to profylaxis with the same aim)

CONTACTS AND LOCATIONS:
Locations (1):
- Östersund Hospital, Östersund, Alberta, Sweden

IPD SHARING:
Plan to Share IPD: No